CLINICAL TRIAL: NCT01346020
Title: Genomic Analysis of Patients With Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: dr. Natalie Put, Department of Human Genetics UZLeuven
Other Study IDs: S53270
Record Dates: First submitted 2011-04-26; First posted 2011-05-02 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- CLL

SUMMARY:
This study aims to characterize clonal evolution in chronic lymphocytic leukemia (CLL) using different approaches and to identify a possible association with disease progression, i.e. therapy initiation.

1. Samples This monocentric study is carried out using representative bioarchived leukemic samples with a diagnosis of CLL, either at diagnosis or at evolution. These bioarchived samples were collected locally at our center during years of diagnostic activity, and were accurately pathologically, cytogenetically and molecularly characterized.
2. Clinical data The clinical data were retrospectively collected through collaboration with the referring physicians.
3. Methods Samples will be investigated by means of (1) conventional cytogenetics, (2) fluorescence in situ hybridization (FISH) and (3) SNP-arrays. After analysis of the array data sets, significant results will be validated and in addition, results will be correlated with clinical data.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CLL,
* at least two available stored samples

Exclusion Criteria:

* at least one inclusion criterium not fulfilled

Ages: 0 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Time to therapy | baseline to day 1 of therapy
  Time from diagnosis to the start of first line therapy

SECONDARY OUTCOMES:
Genetic abnormalities detected by karyotyping, FISH or array-analysis | 13-102 months
  Detection of any type of genetic abnormality or pattern of abnormalities present at diagnosis or at time of disease progression (e.g. median 41 months after diagnosis, range 13-102 months) by means of karyotyping, fluorescent in situ hybridization or array-analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of human genetics, University Hospital Leuven, Leuven, Belgium